CLINICAL TRIAL: NCT01399099
Title: Scar Prevention and the Clinical Effectiveness of a Novel Mechanomodulating Polymer
Brief Title: A Study of a Novel Silicone Dressing to Minimize Scar Formation
Acronym: REFINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neodyne Biosciences, Inc. (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA003; 00016580 (Other Grant/Funding Number: Armed Forces Institute of Regenerative Medicine)
Record Dates: First submitted 2011-06-27; First posted 2011-07-21 (Estimated); Results first posted 2014-12-25 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hypertrophic
Keywords: scar; incision; wound healing; scarring; post-surgical
MeSH Terms: conditions — Hypertrophy; Cicatrix; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- embrace Dressing (Experimental): Investigational Dressing
  Interventions: Device: embrace device
- Standard of Care (No Intervention): Standard of care comparator

INTERVENTIONS:
Device: embrace device — Adhesive bandage/dressing intended to minimize scar formation.
  Other Names: Neodyne Device; embrace dressing; Neodyne Dressing
  Arms: embrace Dressing

SUMMARY:
Neodyne has developed an investigational dressing for post-operative incision care. Neodyne is conducting this research to study whether the investigational dressing, called the Neodyne Dressing, can minimize scar formation in a simple manner.

DETAILED DESCRIPTION:
It is proposed to study a dressing designed to reduce scarring in post-incision skin tissue. It is expected that by managing the incision site during the healing phase, scar formation may be minimized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone a de novo abdominoplasty.
* Appearance of subject's incision is aesthetically similar across length of incision.

Exclusion Criteria:

* Subjects with a history of collagen vascular disease, cutis laxica, connective tissue disease, psoriasis, or lupus.
* Subjects diagnosed with scleroderma.
* Subjects with known adverse reactions to steri-strip tapes, medical tapes, or adhesives.
* Subjects with oozing, dehiscence, non-closed/healed incisions at time of first application.
* Subjects with inability to maintain adequate care of incision.
* Subjects with a body mass index (BMI) > 30.
* Subjects with a weight loss of greater than or equal to 100 lbs within 6 months from date of abdominoplasty.
* Subjects who currently smoke.
* Subjects taking steroid therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney J Rohrich, MD, FACS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (13):
- United States (13):
  - Atherton Plastic Surgery, Atherton, California
  - Vipul R. Dev MD, Bakersfield, California
  - Elite MD, Danville, California
  - Kaufman and Clark Plastic Surgery, Folsom, California
  - The Aesthetic Institute, Fullerton, California
  - The Korman Group, Mountain View, California
  - Newport Plastic Surgery, Newport Beach, California
  - Lauren Greenberg, MD, Palo Alto, California
  - Plastic Surgery Associates of Santa Rose, Santa Rosa, California
  - Joseph Mele, MD, Walnut Creek, California
  - Academy of Clinical Research, Arlington, Texas
  - The University of Texas Southwestern Medical Center - Dept. of Plastic Surgery, Dallas, Texas
  - US Army Institute of Surgical Research, Fort Sam Houston, Texas

REFERENCES:
- [Derived] Longaker MT, Rohrich RJ, Greenberg L, Furnas H, Wald R, Bansal V, Seify H, Tran A, Weston J, Korman JM, Chan R, Kaufman D, Dev VR, Mele JA, Januszyk M, Cowley C, McLaughlin P, Beasley B, Gurtner GC. A randomized controlled trial of the embrace advanced scar therapy device to reduce incisional scar formation. Plast Reconstr Surg. 2014 Sep;134(3):536-546. doi: 10.1097/PRS.0000000000000417. PMID 24804638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Procedures were performed by 12 surgeons at 12 surgery centers between June 2011 and May of 2012.
Groups:
- All Study Participants: Half of the abdominoplasty incision was treated with the embrace device. Half of the abdominoplasty incision was treated according to the investigator's standard of care. Participant served as his own control.
Period: Overall Study
Arm/Group | All Study Participants
Started | 67
6 Months | 47
Completed | 33
Not Completed | 34
Not completed — Lost to Follow-up | 14
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Skin Irritation | 13
Not completed — Infection | 1
Not completed — Miscellaneous | 4

BASELINE CHARACTERISTICS:
Population: After meeting all eligibility criteria, 67 patients were enrolled.
Arm/Group | All Study Participants
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 47
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: Visual Analogue Scale Scar Score (VAS Scar Score) was defined and validated by Duncan et al 2006[1]. This scale consists of a 10cm line representing scar quality, with 0 representing normal skin and 10 indicating a poor scar. The assessor places a mark along the line to represent the appearance of the scar. This mark is translated into a score by measuring its position on the 10cm line to one decimal place. The independent panel used this to scale the primary outcome.
  [1] Duncan J, Bond J, Mason T, Ludlow A, Cridland P, O'Kane S and Ferguson M. Visual Analogue Scale Scoring and Ranking: A Suitable and Sensitive Method for Assessing Scar Quality? Plast. Reconstr. Surg. 118: 909, 2006.
Time Frame: 12 months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treated Side: Half of the abdominoplasty incision was treated with the embrace device.
- Control Side: Half of the abdominoplasty incision was treated according to the Investigator's standard of care. Participant served as his/her own control.
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 33 | 33
score on a scale | 2.90 (1.36) | 3.29 (1.55)

2. Primary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 6 months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treated Side: Half of the abdomnioplasty incision was treated with the embrace device.
- Control Side: Half of the abdomnioplasty incision was treated according to the Investigator's standard of care. Participant served as his/her own control.
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 47 | 47
score on a scale | 3.18 (1.71) | 3.85 (1.77)

3. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - Patient Results
Description: The Patient and Observer Scar Assessment Scale consists of two numeric scales: the Patient Scar Assessment Scale (patient scale) and the Observer Scar Assessment Scale (observer scale). The patient and observer scales have to be completed by the patient and the observer, respectively [1]. The POSAS criteria evaluated by the patients in this study were pain, itching, color, stiffness, thickness, irregularity, and overall opinion. The Patient and Observer Scar Assessment Scale (POSAS) ranges from 1 to 10 with 10 being the worst imaginable or most different.
  [1] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID: 15253184.
Time Frame: 6 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 44 | 44
score on a scale
  Pain | 1.05 (0.21) | 1.21 (0.80)
  Itch | 1.41 (1.24) | 1.52 (1.47)
  Color | 4.75 (2.37) | 5.21 (2.53)
  Stiffness | 2.91 (1.95) | 4.48 (2.60)
  Thickness | 3.34 (2.12) | 4.30 (2.30)
  Irregularity | 3.66 (2.38) | 4.61 (2.64)
  Overall | 3.70 (2.21) | 4.91 (2.75)

4. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - Patient Results
Description: The Patient and Observer Scar Assessment Scale consists of two numeric scales: the Patient Scar Assessment Scale (patient scale) and the Observer Scar Assessment Scale (observer scale). The patient and observer scales have to be completed by the patient and the observer, respectively [1]. The POSAS criteria evaluated by the patients in this study were pain, itching, color, stiffness, thickness, irregularity, and overall opinion.
  [1] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID: 15253184.
Time Frame: 12 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 35 | 35
score on a scale
  Pain | 1.00 (0.00) | 1.06 (0.24)
  Itch | 1.40 (1.24) | 1.29 (1.20)
  Color | 3.80 (2.21) | 4.31 (2.49)
  Stiffness | 2.63 (2.06) | 3.77 (2.43)
  Thickness | 2.86 (2.02) | 3.97 (2.48)
  Irregularity | 3.46 (2.19) | 4.29 (2.58)
  Overall | 3.66 (2.35) | 4.66 (2.80)

5. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - Observer Results
Description: The Patient and Observer Scar Assessment Scale consists of two numeric scales: the Patient Scar Assessment Scale (patient scale) and the Observer Scar Assessment Scale (observer scale). The patient and observer scales have to be completed by the patient and the observer, respectively [1]. The POSAS criteria evaluated by the observers in this study were vascularity, pigmentation, thickness, relief, pliability, surface area, and an overall opinion.
  [1] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID: 15253184.
Time Frame: 6 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 45 | 45
score on a scale
  Vascularity | 2.07 (0.72) | 2.96 (1.46)
  Pigmentation | 2.16 (1.11) | 3.13 (1.58)
  Thickness | 3.07 (2.78) | 3.73 (2.19)
  Relief | 2.78 (1.52) | 3.62 (1.81)
  Pliability | 2.09 (1.00) | 2.98 (1.45)
  Surface Area | 3.07 (2.29) | 3.42 (1.76)
  Overall Opinion | 1.98 (0.62) | 3.02 (1.45)

6. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - Observer Results
Description: as for outcome 5
Time Frame: 12 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 36 | 36
score on a scale
  Vascularity | 1.67 (0.63) | 2.25 (1.18)
  Pigmentation | 1.61 (0.77) | 2.69 (1.98)
  Thickness | 3.36 (3.20) | 3.50 (2.56)
  Relief | 2.56 (1.61) | 3.11 (1.86)
  Pliability | 1.67 (0.68) | 2.25 (1.00)
  Surface Area | 2.92 (2.18) | 2.81 (1.62)
  Overall Opinion | 1.61 (0.55) | 2.50 (1.38)

7. Secondary Outcome: Patient Satisfaction - Scar Minimization
Description: Subjects were were asked to compare the embrace-treated side with the control-treated side with regards to their satisfaction with the scar minimization on their incision.
Time Frame: 6 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 44
Participants
  Very Satisfied | 14
  Satisfied | 18
  Neither Satisfied nor Dissatisfied | 11
  Dissatisfied | 1
  Very Dissatisfied | 0

8. Secondary Outcome: Patient Satisfaction - Recommend
Description: Subjects were were asked to rate how likely they were to recommend embrace treatment to a friend.
Time Frame: 6 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 44
Participants
  Very Likely | 16
  Likely | 19
  Neither likely nor unlikely | 4
  Unlikely | 3
  Very Unlikely | 2

9. Secondary Outcome: Patient Satisfaction - Use Again
Description: Subjects were asked if they were to have another procedure that would leave a scar how likely would they be to use embrace treatment again.
Time Frame: 6 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 44
Participants
  Very likely | 22
  Likely | 10
  Neither likely nor unlikely | 4
  Unlikely | 5
  Very Unlikely | 3

10. Secondary Outcome: Patient Satisfaction - Scar Minimization
Description: as for outcome 7
Time Frame: 12 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 35
Participants
  Very Satisfied | 14
  Satisfied | 11
  Neither Satisfied nor Dissatisfied | 10
  Dissatisfied | 0
  Very Dissatisfied | 0

11. Secondary Outcome: Patient Satisfaction - Recommend
Description: Subjects were were asked to rate how likely they were to recommend embrace treatment to a friend.
Time Frame: 12 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 35
Participants
  Very Likely | 15
  Likely | 11
  Neither Likely nor Unlikely | 5
  Unlikely | 2
  Very Unlikely | 2

12. Secondary Outcome: Patient Satisfaction - Use Again
Description: as for outcome 9
Time Frame: 12 Months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Side
Number analyzed (Participants) | 35
Participants
  Very Likely | 15
  Likely | 12
  Neither Likely nor Unlikely | 3
  Unlikely | 3
  Very Unlikely | 2

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Adverse Events were reported via phone call or in person at weekly site visits for Neodyne dressing applications. Data was collected by investigators on Adverse Event Clinical Report Forms for each participant. After initial 12 weeks of application visits, data was collected at 6 month and 12 month (optional) intervals. Adverse Events data were only collected for the interventional treatment arm.
Groups:
- Treatment Arm: Half of the abdominoplasty incision was treated with the embrace device.
Arm/Group | Treatment Arm | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 40/67 | 40/67
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=67) | All Study Participants (N=67)
Erythema (Skin and subcutaneous tissue disorders) | 7 (11) | 7 (11)
Infection (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (8)
Maceration (Skin and subcutaneous tissue disorders) | 5 (8) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Skin Irritation (Skin and subcutaneous tissue disorders) | 24 (29) | 24 (29)

LIMITATIONS AND CAVEATS:
* The Neodyne Dressing is referred to as the embrace device.
* Grant/Funding source: Armed Forces Institute of Regenerative Medicine is funded by US Army Medical Research and Materiel Command (our collaborator) http://www.afirm.mil/

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No